CLINICAL TRIAL: NCT03312998
Title: Incidence of Metal Failure During First Year Following Transpedicular Screws Fixation of Dorso Lumbar Spine Fracture
Brief Title: Incidence of Metal Failure During First Year Following Transpedicular Screws Fixation of Dorsolumbar Spine Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moh Salah, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17100187
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: SPINAL Fracture
MeSH Terms: conditions — Spinal Fractures | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xrays (Experimental)
  Interventions: Radiation: Xrays

INTERVENTIONS:
Radiation: Xrays — Plain x-rays anteroposterior and lateral views to determine system failure

SUMMARY:
Recording incidence of metal failure in transpedicular screws fixation of dorsal umbra spine fracture during first year follow up

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* post traumatic dorsolumbar spine fracture fixed with short or long segment transpedicular screws
* With or without decompression

Exclusion Criteria:

* pediatric patients
* Pathological fractures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
radiological assessment of transpedicular screws after dorsolumbar fixation | 1 year
  Broken rods screws loosening of screws and nuts

REFERENCES:
- [Background] Riaz-ur-Rehman, Azmatullah, Azam F, Mushtaq, Shah M. Treatment of traumatic unstable thoracolumbar junction fractures with transpedicular screw fixation. J Pak Med Assoc. 2011 Oct;61(10):1005-8. PMID 22356037
- [Background] Wang L, Yan J, Li Y, Xu K, Li S, Tang P, Li H. The influence of hydroxypropyl-beta-cyclodextrin on the solubility, dissolution, cytotoxicity, and binding of riluzole with human serum albumin. J Pharm Biomed Anal. 2016 Jan 5;117:453-63. doi: 10.1016/j.jpba.2015.09.033. Epub 2015 Oct 9. PMID 26454338
- [Background] Moon MS, Kim SS, Lee BJ, Moon JL, Lin JF, Moon YW. Radiographic assessment of congenital C2-3 synostosis. J Orthop Surg (Hong Kong). 2010 Aug;18(2):143-7. doi: 10.1177/230949901001800203. PMID 20808002
- [Background] Moon MS, Choi WT, Sun DH, Chae JW, Ryu JS, Chang H, Lin JF. Instrumented ligamentotaxis and stabilization of compression and burst fractures of dorsolumbar and mid-lumbar spines. Indian J Orthop. 2007 Oct;41(4):346-53. doi: 10.4103/0019-5413.36999. PMID 21139790